CLINICAL TRIAL: NCT02145767
Title: Progesterone for the Prevention of Miscarriage and Preterm Birth in Women With First Trimester Bleeding: PREEMPT Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Haim Abenhaim, Obstetrician & Gynecologist, Maternal Fetal Medicine Specialist, Director of Perinatal Research, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRMT15
Record Dates: First submitted 2014-05-14; First posted 2014-05-23 (Estimated); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Miscarriage; Preterm Birth
MeSH Terms: conditions — Abortion, Spontaneous; Premature Birth | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Progesterone (Experimental): Progesterone 200mg suppository administered vaginally at bedtime until 34 completed weeks of pregnancy.
  Interventions: Drug: Progesterone
- Placebo (Placebo Comparator): Similar appearing suppository containing vehicle alone administered vaginally at bedtime until 34 completed weeks of pregnancy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Progesterone
  Arms: Progesterone
Drug: Placebo
  Arms: Placebo

SUMMARY:
Miscarriages and preterm births are common and serious events affecting women, families, and healthcare systems on many levels. One of the risk factors for miscarriage and preterm birth is bleeding in the first trimester of pregnancy. Progesterone, a hormone that plays a key role during pregnancy, has been proposed as a possible medication to be used in pregnancy to prevent miscarriage and preterm birth among women who have bleeding in their first trimester of pregnancy. Unfortunately, unless sound clinical evidence is obtained through a clinical trial, whether or not progesterone can indeed prevent miscarriage and preterm birth remains uncertain and thus is not a recommended treatment in women with early pregnancy bleeding. The purpose of our study is to evaluate the effect of progesterone for the prevention of miscarriage and preterm birth among women with early pregnancy bleeding. We will carry out a clinical trial in which 850 women will be randomized to receive either progesterone supplementation (425 women) or a similarly appearing placebo (425 women) and the outcome of their pregnancy will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Live intrauterine singleton pregnancy of <14 weeks by crown-rump length on ultrasound with documented fetal cardiac activity
* Presence of a perigestational (subchorionic) hemorrhage on ultrasound

Exclusion Criteria:

* Contraindication to Progesterone
* Any indication for progesterone

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 850 (Estimated)
Dates: Start 2014-12 (Actual); Primary Completion 2021-02 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Miscarriage | From 6-8 weeks of pregnancy until miscarriage
  Occurrence of a miscarriage (<20 weeks)
Preterm birth | From 6-8 weeks of pregnancy until delivery
  Occurrence of preterm birth (<37 weeks)

SECONDARY OUTCOMES:
Maternal outcomes | From 6-8 weeks of pregnancy until 6 weeks post delivery
  Antenatal admissions, treatment of preterm labor etc.
Neonatal outcomes | 2 days to 6 weeks post delivery
  Malformations, growth restriction, prematurity associated morbidity, etc.
Healthcare outcomes | From 6-8 weeks of pregnancy until 6 weeks post delivery
  Hospital costs, etc

CONTACTS AND LOCATIONS:
Overall Officials: Haim Abenhaim, MD, MPH, Principal Investigator — Jewish General Hospital
Locations (7):
- Canada (7):
  - Karma Medical Clinic, Kitchener, Ontario
  - North York General Hospital, North York, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - CHU Sainte-Justine, Montreal, Quebec
  - MUHC Royal Victoria Hospital, Montreal, Quebec
  - St. Mary's Hospital, Montreal, Quebec
  - Hôpital Fleurimont, Sherbrooke, Quebec